CLINICAL TRIAL: NCT01527773
Title: The Obstructive Pulmonary Disease Outcomes Cohort of Switzerland (TOP DOCS): Phenotypes and Vascular Damage in COPD
Brief Title: Phenotypes and Vascular Damage in Chronic Obstructive Pulmonary Disease (COPD)
Acronym: TOPDOCS
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: TOPDOCS V1.2
Record Dates: First submitted 2012-01-18; First posted 2012-02-07 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Cardiovascular disease; Phenotypes
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- COPD cohort: Cohort of patients with proven COPD

SUMMARY:
TOPDOCS is a prospective cohort study including COPD patients from currently six study centers in Switzerland. Patients with COPD GOLD stages I-IV will be enrolled and followed-up annually for at least 3 years. Yearly assessments will include a detailed patient history, quality of life and activity questionnaires, history of exacerbations, lung function, measurements of exercise capacity, measurements of vascular function, exhaled breath analysis and blood sampling. The overall objective of the project is to establish a meticulously characterized cohort of COPD patients living in Switzerland in order to allow high quality research on the pathogenesis, treatment and complications of COPD. The specific aim of the project is to determine clinically relevant COPD phenotypes and biological factors influencing vascular function in COPD patients.

ELIGIBILITY:
Inclusion criteria:

* Proven COPD (GOLD stages I-IV)
* Age: 40-75 years

Exclusion criteria:

* Mental or physical disability precluding informed consent or compliance with the protocol
* Acute or recent (within the last 6 weeks) exacerbation of COPD

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with proven COPD, GOLD stages I-IV
Sampling Method: Non-Probability Sample
Enrollment: 313 (Actual)
Dates: Start 2011-05; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Lung function | The change from baseline in lung function at 3 years
  FEV1

SECONDARY OUTCOMES:
Exacerbations | The number of exacerbations observed within 3 years
  Number of COPD exacerbations observed within 3 years of observation
Cardiovascular risk score | The change from baseline in risk score function at 3 years
  Pocock score
BODE-index | The change from baseline in BODE-index at 3 years
  BODE-Index
Quality of life | The change from baseline in quality of life scale at 3 years
  Quality of life scales
Blood pressure | The change from baseline in mean blood pressure at 3 years
  Mean blood pressure
Activity | The change from baseline in activity at 3 years
  Actigraphy
Hear Arterial Stiffness | The change from baseline in arterial stiffness at 3 years
  Arterial stiffness by pulse wave analysis
Endothelial Function | The change from baseline in endothelial function at 3 years
  Endothelial function assessed by flow-mediated dilatation (FMD)
Exercise capacity | The change from baseline in exercise capacity at 3 years
  6 minute walking test and sit-to-stand test

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Kohler, MD, Principal Investigator — University Hospital Zurich, Division of Pneumology
Locations (1):
- University Hospital Zurich, Pneumology, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Roeder M, Sievi NA, Kohlbrenner D, Clarenbach CF, Kohler M. Arterial Stiffness Increases Over Time in Relation to Lung Diffusion Capacity: A Longitudinal Observation Study in COPD. Int J Chron Obstruct Pulmon Dis. 2020 Jan 23;15:177-187. doi: 10.2147/COPD.S234882. eCollection 2020. PMID 32158204
- [Derived] Sievi NA, Brack T, Brutsche MH, Frey M, Irani S, Leuppi JD, Thurnheer R, Kohler M, Clarenbach CF. "Can do, don't do" are not the lazy ones: a longitudinal study on physical functioning in patients with COPD. Respir Res. 2020 Jan 20;21(1):27. doi: 10.1186/s12931-020-1290-9. PMID 31959169
- [Derived] Sievi NA, Kohler M, Thurnheer R, Leuppi JD, Irani S, Frey M, Brutsche M, Brack T, Clarenbach CF. No impact of exacerbation frequency and severity on the physical activity decline in COPD: a long-term observation. Int J Chron Obstruct Pulmon Dis. 2019 Feb 15;14:431-437. doi: 10.2147/COPD.S188710. eCollection 2019. PMID 30863043
- [Derived] Sievi NA, Brack T, Brutsche MH, Frey M, Irani S, Leuppi JD, Thurnheer R, Kohler M, Clarenbach CF. Physical activity declines in COPD while exercise capacity remains stable: A longitudinal study over 5 years. Respir Med. 2018 Aug;141:1-6. doi: 10.1016/j.rmed.2018.06.013. Epub 2018 Jun 18. PMID 30053953
- [Derived] Clarenbach CF, Sievi NA, Kohler M. Annual progression of endothelial dysfunction in patients with COPD. Respir Med. 2017 Nov;132:15-20. doi: 10.1016/j.rmed.2017.09.005. Epub 2017 Sep 18. PMID 29229089
- [Derived] Sievi NA, Franzen D, Kohler M, Clarenbach CF. Physical inactivity and arterial stiffness in COPD. Int J Chron Obstruct Pulmon Dis. 2015 Sep 10;10:1891-7. doi: 10.2147/COPD.S90943. eCollection 2015. PMID 26392763
- [Derived] Sievi NA, Senn O, Brack T, Brutsche MH, Frey M, Irani S, Leuppi JD, Thurnheer R, Franzen D, Kohler M, Clarenbach CF. Impact of comorbidities on physical activity in COPD. Respirology. 2015 Apr;20(3):413-8. doi: 10.1111/resp.12456. Epub 2015 Jan 6. PMID 25565363
- [Derived] Schonmann M, Sievi NA, Clarenbach CF, Brack T, Brutsche M, Frey M, Irani S, Leuppi JD, Ruediger J, Senn O, Thurnheer R, Kohler M. Physical activity and the frequency of acute exacerbations in patients with chronic obstructive pulmonary disease. Lung. 2015 Feb;193(1):63-70. doi: 10.1007/s00408-014-9673-7. Epub 2014 Dec 13. PMID 25503750